CLINICAL TRIAL: NCT01393704
Title: Vasopressin Administration During Laparoscopic Myomectomy: a Randomized Controlled Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); North Shore Medical Center (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Jon I. Einarsson, Chief, Division of Minimally Invasive Gynecology, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-P-000264/1
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-01

CONDITIONS: Blood Loss, Surgical
Keywords: myomectomy; vasopressin; blood loss
MeSH Terms: conditions — Blood Loss, Surgical; Diabetes Insipidus; Hemorrhage | interventions — Vasopressins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Volume Dilute Vasopressin (Active Comparator): 20 units Vasopressin diluted in 400 mL of Saline, inject 200 mL total of the dilute Vasopressin solution in subserosal location overlying fibroid (total 10 units Vasopressin used).
  Interventions: Drug: Vasopressin
- Low volume dilute vasopressin (Active Comparator): 20 units Vasopressin diluted in 60 mL of Normal Saline, inject 30 mL total of the dilute Vasopressin solution in subserosal location overlying fibroid (total 10 units Vasopressin used).
  Interventions: Drug: Vasopressin

INTERVENTIONS:
Drug: Vasopressin — Dilute vasopressin solution will be injected subserosally into myoma at time of minimally invasive myomectomy.
  Other Names: Pitressin

SUMMARY:
The main purpose of this study is to compare blood loss at the time of laparoscopic or robotically-assisted laparoscopic myomectomy when using different amounts of dilute vasopressin solution. Myomectomy is a surgical procedure to remove fibroids from the uterus. Vasopressin is a synthetic drug used to help decrease blood loss at the time of gynecologic surgery; although very little is know about the optimal dosage and administration.

The investigators plan to perform a randomized clinical trial on patients scheduled for minimally invasive myomectomy. All patients will get the same overall amount of vasopressin. Patients will be assigned by chance to one of two groups: one group will receive higher volume of a more dilute vasopressin solution. The other group will receive a lower volume of a more concentrated solution. The investigators will collect information on operative blood loss and complications related to surgery.

DETAILED DESCRIPTION:
All surgeons who enroll patients into our study are experienced laparoscopic surgeons who have performed at least 100 advanced laparoscopic procedures including hysterectomies and myomectomies. Briefly, our laparoscopic myomectomy technique is as follows: After gaining peritoneal access and placing visual and operative trocars, the surgical site is inspected carefully and fibroid locations identified. After informing the anesthesia team that vasopressin (from pharmaceutical company American Regent 20 units/ml) is about to be injected, the uterus is infiltrated with vasopressin.

Patients will be randomized one of two treatment groups pre-operatively on the day of surgery:

1. One arm will receive injection of 200 ml total of the 0.05 units/ml dilute vasopressin solution (total 10 units Vasopressin used, dilution of 20 units vasopressin in 400 ml of normal saline).
2. The second arm will receive injection of 30 ml total of the 0.3 units/ml dilute vasopressin solution (total 10 units Vasopressin used, dilution of 20 units Vasopressin in 60 mL of Normal Saline).

The procedure is done according to surgeon preference using various energy modalities such as monopolar or Harmonic Scalpel® (Ethicon Endo-Surgery, Cincinnati OH), for making the incision in the uterus. The fibroid is then removed from the uterus and examined. The incision is then closed in several layers with laparoscopic standard suturing technique, and hysterotomy site is generally covered with an adhesion barrier (Gynecare Interceed® (Ethicon Women's Health and Urology, Somerville NJ) or Seprafilm® slurry (Genzyme Biosurgery, Framingham MA)).

Blood Samples:

As per routine, preoperative blood samples to assess hematocrit levels will be taken no greater than 2 weeks prior to surgical date; if no preoperative laboratory studies have been obtained a sample will be drawn on the day of surgery. Postoperative blood samples to assess hematocrit will be taken no sooner than 4 hours after surgery for patients who are discharged the same day; for patients who are monitored overnight in hospital, the lab will be drawn on postoperative day #1.

Follow-up:

Patients will be followed for 8 weeks after surgery to assess for occurrence of any postoperative complication. A member of the team (health care worker such as research assistant who has been trained in HIPPA procedures) will be in charge of abstracting data from the medical records and entering this information into a study database.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for our study include all women who are candidates for a laparoscopic or robotic-assisted laparoscopic myomectomy and are willing to accept randomization.
* The exclusion criteria: for our study include: suspected malignancy or contraindication to morcellation of uterine tissue, history of adverse reaction or allergy to vasopressin, and active cardiovascular or pulmonary disease that would indicate a contradiction to use of vasopressin.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 152 (Actual)
Dates: Start 2011-07; Primary Completion 2015-04 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon I Einarsson, MD,MPH., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham&Women's hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High Volume Dilute Vasopressin | Low Volume Dilute Vasopressin
Started | 76 | 76
Completed | 76 | 76
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Volume Dilute Vasopressin | Low Volume Dilute Vasopressin | Total
Number analyzed (Participants) | 76 | 76 | 152
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 76 | 76 | 152
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.39 (5.68) | 37.87 (7.11) | 37.49 (6.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 76 | 152
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 76 | 76 | 152

OUTCOME MEASURES:

1. Primary Outcome: Estimating Blood Loss at the End of Myomectomy - Hematocrit Percentage
Description: To evaluate whether volume of dilute Vasopressin administered during minimally-invasive myomectomy affects blood loss, three parameters will be collected to assess this outcome. Pre and post-operative hematocrit change (%) was one of these measurement methods.
Time Frame: 5 minutes post-operatively
Population: Due to practice pattern differences among sites, there was some missing data for the change in hematocrit variable, where the hematocrit either pre-operatively or post-operatively was not collected.
Measure: Mean (Standard Deviation); unit: hematocrit percentage
Arm/Group | High Volume Dilute Vasopressin | Low Volume Dilute Vasopressin
Number analyzed (Participants) | 45 | 46
hematocrit percentage | -4.4 (3.9) | -4.0 (3.2)

2. Primary Outcome: Estimating Blood Loss at the End of Myomectomy - Surgeon Estimated Blood Loss
Description: To evaluate whether volume of dilute Vasopressin administered during minimally-invasive myomectomy affects blood loss, three parameters will be collected to assess this outcome: Subjective surgeon's estimate of blood loss (ml) was one measurement method.
Time Frame: 5 minutes post-operatively
Measure: Mean (Standard Deviation); unit: millileters
Arm/Group | High Volume Dilute Vasopressin | Low Volume Dilute Vasopressin
Number analyzed (Participants) | 76 | 76
millileters | 106.2 (3.0) | 119 (3.2)

3. Primary Outcome: Estimating Blood Loss at the End of Myomectomy - Suction Canister Estimated Blood Loss Calculation
Description: To evaluate whether volume of dilute Vasopressin administered during minimally-invasive myomectomy affects blood loss, three parameters will be collected to assess this outcome. Objective calculation of blood loss via the measurement of suction canister fluid (ml) was one of these. The calculation for estimated blood loss will be as follows: EBL = [total suction canister volume] - [volume of irrigation used] - [volume of vasopressin solution injected /2].
Time Frame: 5 minutes post-operatively
Population: Due to practice pattern differences among sites, there was some missing data for suction canister blood loss calculation. In these cases, total suction canister volume and/or volume of irrigation used were not measured.
Measure: Mean (Standard Deviation); unit: millileters
Arm/Group | High Volume Dilute Vasopressin | Low Volume Dilute Vasopressin
Number analyzed (Participants) | 63 | 61
millileters | 178 (265) | 198 (232)

4. Secondary Outcome: Number of Participants With Peri-operative Complications
Description: Intra or post-operative complications (including but not limited to need for blood transfusion or adverse effect related to Vasopressin).
Time Frame: 8 weeks postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | High Volume Dilute Vasopressin | Low Volume Dilute Vasopressin
Number analyzed (Participants) | 76 | 76
Participants | 9 | 10

5. Secondary Outcome: Total Operation Time
Description: Time from incision to end of surgery
Time Frame: 5 minutes postoperatively
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | High Volume Dilute Vasopressin | Low Volume Dilute Vasopressin
Number analyzed (Participants) | 76 | 76
minutes | 176.8 (82.09) | 165.5 (70.26)

ADVERSE EVENTS:
Time Frame: Adverse events data was collected for a period of 4 years, from the start of the study (July 2011), to completion of the study (June 2015). The time frame for reporting adverse events will be within 7 calendar days of the adverse event. Patients were assessed from the time of their initial consult to 8 weeks following surgery.
Description: If an adverse event occurs to any patients enrolled in this study, the primary investigator will conduct an investigation to determine if the event was related to the study protocol (ie: administration of vasopressin). If the event is clearly linked, or insufficient data exists to determine relationship of event to study protocol, then the investigator will report the event to the IRB. Any protocol-related complication will be communicated to investigators at other sites as well.
Arm/Group | High Volume Dilute Vasopressin | Low Volume Dilute Vasopressin
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/76
Other Adverse Events (participants affected / at risk) | 0/76 | 0/76

LIMITATIONS AND CAVEATS:
Due to practice pattern differences among sites, there was some missing data for the change in hematocrit variable, and a smaller amount of data missing for suction canister blood loss calculation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes